CLINICAL TRIAL: NCT01113320
Title: A Double-blind, Randomized, Placebo-controlled, Parallel-group, Dose Escalation Trial to Explore the Potential Antidyskinetic Properties of Safinamide in Patients With Parkinson's Disease Suffering From Levodopa Induced Dyskinesias
Brief Title: Safinamide in Levodopa Induced Dyskinesia in Parkinson's Disease Subjects
Acronym: Safinamide-LID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Newron Pharmaceuticals SPA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: EMR701165_023
Record Dates: First submitted 2010-04-08; First posted 2010-04-29 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2012-01

CONDITIONS: Parkinson's Disease
Keywords: Safinamide - Parkinson's disease - Levodopa induced dyskinesia; Advanced idiopathic PD patients treated with L-dopa and suffering from temporally predictable L-dopa induced peak-dose dyskinesia.
MeSH Terms: conditions — Parkinson Disease | interventions — safinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Safinamide (Active Comparator)
  Interventions: Drug: Safinamide

INTERVENTIONS:
Drug: Placebo — Evaluable dose levels are 100 mg (8 days), 200 mg (10 days), and 300 mg (42 days). Intermediate dose levels are 150 mg (Study days 9-11) and 250 mg (Study days 23-25) and have a duration of three days. Safinamide and identical Placebo will be provided in tablets equivalent of 50 mg in blisters. Dosing will be achieved using appropriate multiples of these tablet strengths
  Arms: Placebo
Drug: Safinamide — Evaluable dose levels are 100 mg (8 days), 200 mg (10 days), and 300 mg (42 days). Intermediate dose levels are 150 mg (Study days 9-11) and 250 mg (Study days 23-25) and have a duration of three days. Safinamide will be provided in tablets of 50 mg in blisters. Dosing will be achieved using appropriate multiples of these tablet strengths
  Arms: Safinamide

SUMMARY:
Approximately twenty four (24) subjects will participate in this research trial. The research trial will be conducted in approximately twelve (12) medical centers in the following countries: Germany, France, South Africa, Austria and Canada. The research trial will last until December 2011.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has given his/her written informed consent to participate in the trial.
2. The subject presents with a diagnosis of idiopathic Parkinson's disease according to the United Kingdom (UK) Parkinson's Disease Society Brain Bank Clinical Diagnosis Criteria
3. The subject is an out-patient aged 30 years or above.
4. PD subjects with a Hoehn and Yahr disease staging of II-IV (in the ON state).
5. PD subjects experiencing levodopa induced dyskinesias, specifically predictable peak-dose dyskinesia.
6. Peak-dose dyskinesia must be considered by the subject to be problematic and/or disabling.
7. Peak-dose dyskinesia must warrant medical treatment in the Investigator's opinion.
8. The subject has participated successfully in a diary-card training session.
9. In the judgment of the Investigator based on the subject's history, previous treatments, and the clinical presentation, the subject is considered as being optimally treated at screening (i.e., further adjustments of current medication will not further improve the subject's symptoms of Parkinson's disease).
10. Stable dose of PD drugs for at least 4 weeks before Screening Visit. This may include: levodopa dopamine agonists, c-ortho methyl transferase (COMT) inhibitors, and anticholinergics.
11. The dose of levodopa and all PD drugs used during the trial must remain unchanged throughout the trial.
12. Female subjects must be neither pregnant or breast-feeding and must lack child-bearing potential, as defined either by:

    1. be either post menopausal for at least 2 years , surgically sterilised or have undergone hysterectomy, or
    2. if of child bearing potential, be willing to avoid pregnancy by using an adequate method of contraception for four weeks prior to, during and four weeks after the last dose of trial medication. For the purposes of this trial, women of childbearing potential are defined as all female subjects after puberty unless they are post-menopausal for at least two years, are surgically sterile or are sexually inactive.
13. The subject shows adequate compliance with the schedule for intake of trial medication and the completion of the diaries.

Exclusion Criteria:

1. The subject has participated in any safinamide clinical trial before.
2. The subject is experiencing exclusively diphasic, off state, myoclonic, dystonic, or akathetic dyskinesias without peak dose dyskinesia.
3. (For female subjects) The subject is pregnant or lactating.
4. Treatment with a MAO-B inhibitor within the eight weeks prior to the screening visit.
5. Treatment with amantadine in the four weeks prior to the screening visit or budipine in the eight weeks prior to the screening visit.
6. Treatment with opioids (e.g., tramadol, meperidine derivatives), serotonin norepinephrine reuptake inhibitors (SNRIs) (e.g. venlafaxine, duloxetine), tri- or tetra-cyclic antidepressants, in the past 8 weeks prior to the screening visit. Dextromethorphan will be permitted if used for treating cough.
7. The subject has received neurosurgical intervention related to PD (e.g. deep brain stimulation, thalamotomy etc.) or is scheduled to do so during the trial period.
8. Current clinically significant gastro-intestinal, renal, hepatic, endocrine, pulmonary or cardiovascular disease, including acute gastric ulcer, hypertension that is not well controlled, asthma, chronic obstructive pulmonary disease (COPD), and unstable Type I diabetes. Subjects with a history of gastric ulcer who have not had a recent episode of acute gastritis and are not currently experiencing gastric pain will be eligible for inclusion.
9. Neoplastic disorder, which is either currently active or has been in remission for less than one year.
10. Diagnosis of HIV, or positive test for Hepatitis C antibodies, or Hepatitis B surface antigen.
11. Concomitant disease likely to interfere with trial medication (e.g. capable of altering absorption, metabolism, or elimination of the trial drug).
12. The subject has any clinically significant illness that, in the Investigator's opinion, might interfere with the subject's ability to participate in the trial.
13. Second- or third-degree atrio-ventricular block or sick sinus syndrome, uncontrolled atrial fibrillation, severe or unstable angina, congestive heart failure, myocardial infarction within 3 months of the screening visit, or a significant ECG abnormality, including corrected QT interval (QTc) - 450 msec (males) or - 470 msec (females), where QTc is based on Bazett's correction method.
14. Ophthalmologic history including any of the following conditions: albino subjects, family history of hereditary retinal disease, progressive and/or severe diminution of visual acuity (i.e., 20/70), retinitis pigmentosa, retinal pigmentation due to any cause, any active retinopathy or ocular inflammation (uveitis), or diabetic retinopathy
15. The subject is suffering from any dementia or other psychiatric illness that prevents him/her from giving informed consent, i.e. Montreal Cognitive Assessment (MoCA) <23 points.
16. Signs and symptoms suggestive of transmissible spongiform encephalopathy, or family members who suffer(ed) from such.
17. Known hypersensitivity to the trial treatment(s), including placebo or other comparator drug(s).
18. The subject has legal incapacity or limited legal capacity.
19. The subject is participating in another clinical trial or has done so within the past 30 days
20. Treatment with a drug that has hepatotoxic potential, e.g., tamoxifen, within 4 weeks, or received radiation therapy or a drug with cytotoxic potential, e.g, chemotherapy, within one year prior to the screening visit.
21. Subjects with current diagnosis of substance abuse (DSM-IV) or history of alcohol or drug abuse in the past three months.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-04; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The maximum reduction in Unified Dyskinesia Rating Score (UDysRS) compared to baseline across all post-baseline dose visits. | Day 66

SECONDARY OUTCOMES:
Complete new Movement Disorder Society - Unified Parkinson Disease Rating Scale (MDS-UPDRS) and subscales | At each individual post-dose visit: Baseline
Complete new Movement Disorder Society - Unified Parkinson Disease Rating Scale (MDS-UPDRS) and subscales | At each individual post-dose visit: Day 8
Complete new Movement Disorder Society - Unified Parkinson Disease Rating Scale (MDS-UPDRS) and subscales | At each individual post-dose visit: Day 22
Complete new Movement Disorder Society - Unified Parkinson Disease Rating Scale (MDS-UPDRS) and subscales | At each individual post-dose visit: Day 36
Complete new Movement Disorder Society - Unified Parkinson Disease Rating Scale (MDS-UPDRS) and subscales | At each individual post-dose visit: Day 66
Complete new Movement Disorder Society - Unified Parkinson Disease Rating Scale (MDS-UPDRS) and subscales | At each individual post-dose visit: Day 101
Unified Dyskinesia Rating Scale (UDysRS) and subscales (historical and objective) | At each individual visit: Baseline
Unified Dyskinesia Rating Scale (UDysRS) and subscales (historical and objective) | At each individual visit: Day 8
Unified Dyskinesia Rating Scale (UDysRS) and subscales (historical and objective) | At each individual visit: Day 22
Unified Dyskinesia Rating Scale (UDysRS) and subscales (historical and objective) | At each individual visit: Day 36
Unified Dyskinesia Rating Scale (UDysRS) and subscales (historical and objective) | At each individual visit: Day 66
Unified Dyskinesia Rating Scale (UDysRS) and subscales (historical and objective) | At each individual visit: Day 101
Patient's diary (Hauser diary, all parts) | At each trial visit: Baseline
  Hauser patient diary: daily total "on" time (ON w/o dyskinesia, or ON with non-troublesome dyskinesia), and daily total "off" time as measured by the patients' diary over the study period.
Patient's diary (Hauser diary, all parts) | At each trial visit: Day 8
  Hauser patient diary: daily total "on" time (ON w/o dyskinesia, or ON with non-troublesome dyskinesia), and daily total "off" time as measured by the patients' diary over the study period.
Patient's diary (Hauser diary, all parts) | At each trial visit: Day 22
  Hauser patient diary: daily total "on" time (ON w/o dyskinesia, or ON with non-troublesome dyskinesia), and daily total "off" time as measured by the patients' diary over the study period.
Patient's diary (Hauser diary, all parts) | At each trial visit: Day 36
  Hauser patient diary: daily total "on" time (ON w/o dyskinesia, or ON with non-troublesome dyskinesia), and daily total "off" time as measured by the patients' diary over the study period.
Patient's diary (Hauser diary, all parts) | At each trial visit: Day 66
  Hauser patient diary: daily total "on" time (ON w/o dyskinesia, or ON with non-troublesome dyskinesia), and daily total "off" time as measured by the patients' diary over the study period.
Patient's diary (Hauser diary, all parts) | At each trial visit: Day 101
  Hauser patient diary: daily total "on" time (ON w/o dyskinesia, or ON with non-troublesome dyskinesia), and daily total "off" time as measured by the patients' diary over the study period.
Parkinson's Disease Dyskinesia Scale (PDYS-26) (dyskinesia specific Activities of Daily Living (ADL) questionnaire) | At each trial visit: Baseline
Parkinson's Disease Dyskinesia Scale (PDYS-26) (dyskinesia specific Activities of Daily Living (ADL) questionnaire) | At each trial visit: Day 8
Parkinson's Disease Dyskinesia Scale (PDYS-26) (dyskinesia specific Activities of Daily Living (ADL) questionnaire) | At each trial visit: Day 22
Parkinson's Disease Dyskinesia Scale (PDYS-26) (dyskinesia specific Activities of Daily Living (ADL) questionnaire) | At each trial visit: Day 36
Parkinson's Disease Dyskinesia Scale (PDYS-26) (dyskinesia specific Activities of Daily Living (ADL) questionnaire) | At each trial visit: Day 66
Parkinson's Disease Dyskinesia Scale (PDYS-26) (dyskinesia specific Activities of Daily Living (ADL) questionnaire) | At each trial visit: Day 101
Clinical Global Impression (CGI) (dyskinesia specific) | At each trial visit: Baseline
  Scales measure the overall impression both the investigator and the patient have about the subject's general health. This is measured at baseline and the impression of change versus is measured at each visit. Here we are measuring efficacy.
Clinical Global Impression (CGI) (dyskinesia specific) | At each trial visit: Day 8
  Scales measure the overall impression both the investigator and the patient have about the subject's general health. This is measured at baseline and the impression of change versus is measured at each visit. Here we are measuring efficacy.
Clinical Global Impression (CGI) (dyskinesia specific) | At each trial visit: Day 22
  Scales measure the overall impression both the investigator and the patient have about the subject's general health. This is measured at baseline and the impression of change versus is measured at each visit. Here we are measuring efficacy.
Clinical Global Impression (CGI) (dyskinesia specific) | At each trial visit: Day 36
  Scales measure the overall impression both the investigator and the patient have about the subject's general health. This is measured at baseline and the impression of change versus is measured at each visit. Here we are measuring efficacy.
Clinical Global Impression (CGI) (dyskinesia specific) | At each trial visit: Day 66
  Scales measure the overall impression both the investigator and the patient have about the subject's general health. This is measured at baseline and the impression of change versus is measured at each visit. Here we are measuring efficacy.
Clinical Global Impression (CGI) (dyskinesia specific) | At each trial visit: Day 101
  Scales measure the overall impression both the investigator and the patient have about the subject's general health. This is measured at baseline and the impression of change versus is measured at each visit. Here we are measuring efficacy.
Patient Global Impression (PGI) (dyskinesia specific) | At each trial visit: Baseline
  Scales measure the overall impression both the investigator and the patient have about the subject's general health. This is measured at baseline and the impression of change versus is measured at each visit. Here we are measuring efficacy.
Patient Global Impression (PGI) (dyskinesia specific) | At each trial visit: Day 8
  Scales measure the overall impression both the investigator and the patient have about the subject's general health. This is measured at baseline and the impression of change versus is measured at each visit. Here we are measuring efficacy.
Patient Global Impression (PGI) (dyskinesia specific) | At each trial visit: Day 22
  Scales measure the overall impression both the investigator and the patient have about the subject's general health. This is measured at baseline and the impression of change versus is measured at each visit. Here we are measuring efficacy.
Patient Global Impression (PGI) (dyskinesia specific) | At each trial visit: Day 36
  Scales measure the overall impression both the investigator and the patient have about the subject's general health. This is measured at baseline and the impression of change versus is measured at each visit. Here we are measuring efficacy.
Patient Global Impression (PGI) (dyskinesia specific) | At each trial visit: Day 66
  Scales measure the overall impression both the investigator and the patient have about the subject's general health. This is measured at baseline and the impression of change versus is measured at each visit. Here we are measuring efficacy.
Patient Global Impression (PGI) (dyskinesia specific) | At each trial visit: Day 101
  Scales measure the overall impression both the investigator and the patient have about the subject's general health. This is measured at baseline and the impression of change versus is measured at each visit. Here we are measuring efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Willmer, MD, Study Director — Merck Serono S.A., Geneva
Locations (11):
- Austria (2):
  - Medical University Graz, Klinische Abteilung für Spezielle Neurologie, Graz
  - Medical University Innsbruck, Dept. of Neurology, Innsbruck
- Quebec Memory and Motor Skills Disorders, Québec, Canada
- France (2):
  - Hôpital Roger Sallengro, Lille
  - CIC-Hospital Purpan, Toulouse
- Germany (3):
  - Neurologie Berlin Praxen, Berlin
  - St. Josef Hospital, Klinik für Neurologie, Bochum
  - Facharzt für Neurologie und Psychiatrie, Düsseldorf
- South Africa (3):
  - Medical and Dental center (ZAF), Johannesburg
  - Sunninghill Hospital, Johannesburg
  - Willows Medical Centre, Pretoria